CLINICAL TRIAL: NCT05936034
Title: Comparative Study of the Quality of Life of Patients Suffering From OTOTOXICITY Due to Chemotherapy Based on Platinum Salts Fitted With a Hearing Aid Compared to Those Not Fitted.
Acronym: PROTOTOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02141-44
Record Dates: First submitted 2023-06-21; First posted 2023-07-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Ototoxicity, Drug-Induced; Quality of Life; Hearing Disorders
MeSH Terms: conditions — Neoplasms; Ototoxicity; Hearing Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients suffering from chemotherapy-induced ototoxicity (Active Comparator): Arm 1: Patients with chemotherapy-induced ototoxicity who continue their usual care.
  Interventions: Other: Patients suffering from chemotherapy-induced ototoxicity
- Patients suffring from chemotherapy-induced ototoxicity wearing hearing aids (Experimental): Arm 2: Experimental group patients with chemotherapy-induced ototoxicity wearing a hearing aid to evaluate quality of life.
  Interventions: Other: Patients suffring from chemotherapy-induced ototoxicity wearing hearing aids

INTERVENTIONS:
Other: Patients suffering from chemotherapy-induced ototoxicity — At baseline,
  * medical staff carries out a clinical and audiometric and/or tintometric examination
  * patient completes the SF36 survey (36 Item Short-Form Health Survey)
  * Patients will then be randomized to either:
    * Control group: standard support; Once the patient has been fit, he continues his carcinological treatment with platinum-based chemotherapy according to the recommendations specific to his pathology.
  At one, three and six months after fitting,
  * medical staff carries out a clinical examination
  * This visit will be scheduled when the patient arrives as part of their standard care. all patients included in the study will have a clinical examination and an audiometric and/or tinnitus examination and should complete an SF36 quality of life questionnaire.
  Only at the last visit (6 months) all patients included should complete a satisfaction questionnaire.
  Arms: Patients suffering from chemotherapy-induced ototoxicity
Other: Patients suffring from chemotherapy-induced ototoxicity wearing hearing aids — At baseline,
  * medical staff carries out a clinical and audiometric and/or tintometric examination
  * patient completes the SF36 survey (36 Item Short-Form Health Survey)
  * Patients will then be randomized to either:
    * Experimental group: standard treatment with hearing aids (wearing a hearing aid).
  Once the patient has been fit, he continues his carcinological treatment with platinum-based chemotherapy according to the recommendations specific to his pathology.
  At one, three and six months after fitting,
  * medical staff carries out a clinical examination
  * This visit will be scheduled when the patient arrives as part of their standard care. all patients included in the study will have a clinical examination and an audiometric and/or tinnitus examination and should complete an SF36 quality of life questionnaire.
  Only at the last visit (6 months) all patients included should complete a satisfaction questionnaire.
  Arms: Patients suffring from chemotherapy-induced ototoxicity wearing hearing aids

SUMMARY:
There are many undesirable effects associated with platinum-based cancer treatments (renal failure, anaemia, etc.). Their administration also leads to neurosensory problems such as ototoxicity, tinnitus and reduced hearing acuity. According to a the French survey (2018), 39.7% of people suffer from hearing problems due to cancer treatments, five years after a cancer diagnosis.

Improving side effects such as hypoacusis and tinnitus can significantly improve patients' quality of life and adherence to treatment. Many clinical trials proposed a medicinal solution to patients receiving platinum-based cancer treatments but none has led to a consensus on management.

The aim of the study is to offer patients receiving platinum-based chemotherapy and suffering from hearing problems a hearing aid to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient currently undergoing treatment with platinum-based chemotherapy and suffering from hypoacusia consistent with the treatment or presenting a worsening of already existing hypoacusis consistent with the start of treatment with platinum-based chemotherapy
* Patient whose hypoacusis is confirmed by the audiometric test
* Patient able and willing to follow all study procedures in accordance with the protocol.
* Patient having understood, signed and dated the consent form
* Patient affiliated to the social security system

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Persons deprived of liberty or under guardianship (including curatorship)
* Impossibility of submitting to medical monitoring of the trial for geographical, social or psychological reasons
* Patient with a contraindication to wearing hearing aids
* Patient already fitted
* Patient already included in a protocol including an experimental molecule
* Patient who has not started treatment with platinum-based chemotherapy
* Patient presenting only tinnitus without hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2027-09-04 (Estimated); Study Completion 2028-07-04 (Estimated)

PRIMARY OUTCOMES:
Quality of life of patients | 6 months
  The quality of life of patients with hearing aids suffering from ototoxicity due to platinum-based chemotherapy will be assessed using the 36 Item Short-Form Health Survey (SF36).
  [score 0 to 100 : score 0 representing the lowest possible scores and score 100 representing the highest possible scores. A higher score means better health.

SECONDARY OUTCOMES:
Measuring hearing and the onset of tinnitus in patients | 6 months
  Hearing and the onset of tinnitus in hearing-aided patients suffering from chemotherapy-induced ototoxicity will be assessed by Hertz/Decibel measurement using an audiometer
Patient compliance to wearing a hearing aid | 6 months
  Hearing aid compliance will be assessed according to the proportion of patients completing 6-month follow-up with a hearing aid among all included patients.

CONTACTS AND LOCATIONS:
Overall Officials: ROMINA MASTRONICOLA, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No